CLINICAL TRIAL: NCT03044977
Title: Phase 1 Trial Using 131I MIBG and 90Y DOTATOC in a Dosimetrically Determined Optimal Combination for Therapy of Selected Patients With Midgut Neuroendocrine Tumors.
Brief Title: Study to Evaluate the Safety of Combining Two Radionuclide Therapies to Treat Mid-gut Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: David Bushnell (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Holden Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, David Bushnell, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201608857; P50CA174521-02 (NIH)
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Neuroendocrine Tumor, Malignant; Neuroendocrine Tumor Gastrointestinal, Hormone-Secreting
Keywords: 3-Iodobenzylguanidine; dose-response relationship, radiation; theranostic; radionuclide; MIBG; DOTA
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 90Y-octreotide, DOTA-Tyr(3)-; 3-Iodobenzylguanidine

STUDY DESIGN:
Intervention Model Description: dose-escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): This is the initial treatment arm. 131I-MIBG and 90Y-DOTATOC are administered once per cycle, for up to 2 cycles 12 weeks apart.
  Radiation exposure to the bone marrow is limited to 150 centiGray (cGy) Radiation exposure to the kidneys is limited to 1900 centiGray (cGy)
  Interventions: Drug: 90Y-DOTA-3-Tyr-Octreotide; Drug: 131I-MIBG
- Cohort 2 (Experimental): This treatment arm is opened if Cohort 1 is successful. 131I-MIBG and 90Y-DOTATOC are administered once per cycle, for up to 2 cycles 12 weeks apart.
  Radiation exposure to the bone marrow is limited to 200 centiGray (cGy) Radiation exposure to the kidneys is limited to 2300 centiGray (cGy)
  Interventions: Drug: 90Y-DOTA-3-Tyr-Octreotide; Drug: 131I-MIBG
- Cohort 3 (Experimental): This treatment arm is opened if Cohort 2 is successful. 131I-MIBG and 90Y-DOTATOC are administered once per cycle, for up to 2 cycles 12 weeks apart.
  Radiation exposure to the bone marrow is limited to 250 centiGray (cGy) Radiation exposure to the kidneys is limited to 2300 centiGray (cGy)
  Interventions: Drug: 90Y-DOTA-3-Tyr-Octreotide; Drug: 131I-MIBG
- Cohort -1 (alternative cohort) (Experimental): This treatment arm is opened if Cohort 1 is not tolerated.
  131I-MIBG and 90Y-DOTATOC are administered once per cycle, for up to 2 cycles 12 weeks apart.
  Radiation exposure to the bone marrow is limited to 100 centiGray (cGy) Radiation exposure to the kidneys is limited to 1500 centiGray (cGy)
  No further dose evaluations are done after this cohort is completed.
  Interventions: Drug: 90Y-DOTA-3-Tyr-Octreotide; Drug: 131I-MIBG
- Cohort 2.1 (renal alternative) (Experimental): This treatment arm is opened if the kidney radiation exposure was not tolerated in cohort 2.
  131I-MIBG and 90Y-DOTATOC are administered once per cycle, for up to 2 cycles 12 weeks apart.
  Radiation exposure to the bone marrow is limited to 200 centiGray (cGy) Radiation exposure to the kidneys is limited to 1500 centiGray (cGy)
  No further dose evaluations are done after this cohort is completed.
  Interventions: Drug: 90Y-DOTA-3-Tyr-Octreotide; Drug: 131I-MIBG
- Cohort 2.2 (bone marrow alternative) (Experimental): This treatment arm is opened if the kidney radiation exposure was not tolerated in cohort 2.
  131I-MIBG and 90Y-DOTATOC are administered once per cycle, for up to 2 cycles 12 weeks apart.
  Radiation exposure to the bone marrow is limited to 100 centiGray (cGy) Radiation exposure to the kidneys is limited to 2300 centiGray (cGy)
  No further dose evaluations are done after this cohort is completed.
  Interventions: Drug: 90Y-DOTA-3-Tyr-Octreotide; Drug: 131I-MIBG
- Cohort 3.1 (renal alternative) (Experimental): This treatment arm is opened if the kidney radiation exposure was not tolerated in cohort 3.
  131I-MIBG and 90Y-DOTATOC are administered once per cycle, for up to 2 cycles 12 weeks apart.
  Radiation exposure to the bone marrow is limited to 250 centiGray (cGy) Radiation exposure to the kidneys is limited to 1900 centiGray (cGy)
  No further dose evaluations are done after this cohort is completed.
  Interventions: Drug: 90Y-DOTA-3-Tyr-Octreotide; Drug: 131I-MIBG
- Cohort 3.2 (bone marrow alternative) (Experimental): This treatment arm is opened if the kidney radiation exposure was not tolerated in cohort 2.
  131I-MIBG and 90Y-DOTATOC are administered once per cycle, for up to 2 cycles 12 weeks apart.
  Radiation exposure to the bone marrow is limited to 150 centiGray (cGy) Radiation exposure to the kidneys is limited to 2300 centiGray (cGy)
  No further dose evaluations are done after this cohort is completed.
  Interventions: Drug: 90Y-DOTA-3-Tyr-Octreotide; Drug: 131I-MIBG

INTERVENTIONS:
Drug: 90Y-DOTA-3-Tyr-Octreotide — Peptide receptor radiotherapy (PRRT) using Yttrium-90 as the active radionuclide. For intravenous administration only.
  Other Names: 90Y DOTATOC
Drug: 131I-MIBG — Peptide receptor radiotherapy (PRRT) using Iodine-131 as the active radionuclide. For intravenous administration only.

SUMMARY:
This study is designed to identify the best tolerated doses of [131]Iodine-MIBG and [90]Yttrium-DOTATOC when co-administered to treat midgut neuroendocrine tumors. These drugs (131I-MIBG, 90Y-DOTATOC) are radioactive drugs, known as radionuclide therapy. Currently, the safest and best tolerated doses of these drugs (when combined together) is unknown.

DETAILED DESCRIPTION:
[131]Iodine-MIBG and [90]Yttrium-DOTATOC are radioactive drugs designed to treat specific tumor cells. These drugs are a combination of the radiation (131-Iodine, 90-Yttrium) and a protein that targets the tumor cell (MIBG or DOTATOC). Because these proteins are attracted to, and stick to, the tumor, the radiation is centered in the tumors. This kills more tumor cells and minimizes radiation-damage to healthy tissues, like the heart and lungs.

Two organs still absorb some of the radiation, though: bone marrow and the kidney. These organs limit how much radiation can be given to tumors, but we don't know how much radiation is too much. Too much radiation to bone marrow can result in anemia. Too much radiation to the kidneys can result in kidney failure. From prior radiation therapies, we have a general idea of how much radiation we can give safely.

131I-MIBG and 90Y-DOTATOC have never been given together. We want to give them together because many times, tumors are actually groups of different types of cells. This means, not all the cells respond to therapy the same way. If some tumor cells survive therapy, the tumor will continue to grow and eventually come back. We know some mid-gut neuroendocrine tumors (NETs) have targets for DOTATOC and some other mid-gut NETs have targets for MIBG. We also have now identified that some people with mid-gut NETs have different tumors: some with targets for MIBG and some with targets for DOTATOC. For these people, this means treating only with 131I-MIBG or 90Y-DOTATOC will not be enough to treat their cancer. They need both radioactive drugs.

Because we are combining these radioactive drugs, this study is known as a first-in-man study. We are also using a special imaging to help us estimate the radiation dose to the bone marrow and to the kidneys. This is what decides the final dose of 131I-MIBG and 90Y-DOTATOC.

Before receiving therapy, participants will be asked to undergo imaging to verify they have both MIBG and DOTATOC tumor types:

* participants are given very small doses of radioactive drugs
* a special camera (SPECT/CT) collects images (scans)
* imaging (scans) are done over 3 calendar days
* blood samples are taken at that time, too, to measure the circulating amount of tracer doses

If the scans show a participant has both MIBG and DOTATOC tumors, therapy is given:

* a customized dose of 90Y-DOTATOC is given on day 1 of a treatment cycle. This is given outpatient.
* a customized dose of 131I-MIBG is given on day 2 of a treatment cycle. This is given inpatient (admitted to the hospital).
* participants are monitored through blood tests to identify the side effects of therapy.

Each participant can have up to 2 cycles of therapy. The cycles are 12 weeks apart.

The doses for 90Y-DOTATOC and 131I-MIBG are decided based on radiation to the bone marrow and radiation to the kidney. Doses are decided by how well other participants have done on this study.

Participants have life long follow-up for this study. This is very important, because a study like this has not been done.

ELIGIBILITY:
A 2-step eligibility is utilized for this study.

STEP 1:

Inclusion Criteria:

* Ability to understand and the willingness to provide informed consent.
* A pathologically confirmed (histology or cytology) malignant neoplasm that is determined to be well-differentiated neuroendocrine tumor (i.e. grade 1 or grade 2). The primary tumor location should be known or believed to be midgut, or pheochromocytoma, or paraganglioma.
* Disease not amenable to curative intent treatment (primarily surgery) and in addition has shown either clinical or radiographic progression on all available (non-radionuclidic) therapies known to confer clinical benefit.
* SSTR positive sites as demonstrated by either SSTR2 positivity (2+ or 3+ intensity and greater than 10% tumor cell occupying the receptors) or a nuclear medicine scan utilizing 111In-DTPA-Phe3-Octreotide (Octreoscan™) or 68Ga-DOTA-tyr3-Octreotide within 12 months prior to anticipated C1D1 demonstrating SSTR positive tumor sites
* ≥1 tumor site must have demonstrated uptake equal to or greater than normal liver as documented by nuclear scan imaging
* ≥1 evaluable site of disease measuring ≥ 1.5 cm in diameter on CT or MRI as measured per RECIST
* ≥ 18 to 70 years at the time of study drug administration.
* Karnofsky Performance Status at least 70%
* Agrees to contraception.

Exclusion criteria:

* Patients who are considered a fall risk.
* Women who are pregnant or breast feeding.
* Surgery, radiation or chemotherapy within 4 weeks of proposed step 1 start date.
* Prior peptide-receptor radiotherapy (PRRT).
* Investigational drug within 4 weeks of proposed step 1 start date.
* More than one concurrent, malignant disease.
* History of congestive heart failure and cardiac ejection fraction ≤ 40%.
* Patients for whom, in the opinion of their physician, a 24-hour discontinuation of somatostatin analogue therapy represents a health risk.
* Patients who are unable to discontinue medications known to affect MIBG uptake
* Proteinuria, grade 2 (i.e., ≥ 2+proteinuria).
* Long-acting somatostatin analogue treatment within 14 days of proposed step 1 start date.
* Prior external beam radiation involving kidneys (scatter doses of < 500 cGy to a single kidney or radiation to < 50% of a single kidney is acceptable).
* Prior external beam radiation (including brachytherapy) involving 25% of bone marrow (excluding scatter doses of ≤ 5 Gy).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 90Y-DOTA-tyr3-Octreotide, Octreoscan®, 68Ga-Octreotide, or 131I-MIBG.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

If a subject meets STEP 1 criteria, a serial SPECT scan is performed for dosimetry. Step 2 criteria must be met and verified prior to therapy initiation.

STEP 2:

Inclusion Criteria:

* Subjects must demonstrate at least one of the following:

  * One or more MIBG+ and DOTATOC- tumors in addition to one or more DOTATOC+ tumors, and/or,
  * One or more tumor sites where the calculated "safe" radiation tumor dose is higher by at least 25% with a combination of 131I-MIBG and 90Y-DOTATOC than it is with 90Y DOTATOC alone, or,
* Within 2 weeks of study drug administration for therapeutic intent, patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥ 2000 cells/mm3
  * platelets ≥100,000 cells/mm3
  * total bilirubin <1.5 x institutional ULN for age and weight
  * AST(SGOT) ≤ 2.5 x institutional ULN
  * ALT (SGPT) ≤ 2.5 x institutional ULN
  * eGFR ≥ 50 mL/min/1.73 m2 (Cockroft Gault formula)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
glomular filtration rate (eGFR) | 4 and 8 weeks after each treatment, then at 3, 6, & 9 months after the last treatment
  Evaluate renal toxicity using eGFR measurement
urine protein | Monthly beginning 4 weeks after the first treatment through 6 months after the last treatment
  Evaluate renal toxicity using urine protein measurement
platelet count decreased | Weeks 4, 5, 6, 7, 8 after each therapy and then 3, 6, & 12 months after the last treatment
  Evaluate bone marrow toxicity using platelet counts
absolute neutrophil count decreased | Weeks 4, 5, 6, 7, 8 after each therapy and then 3, 6, & 12 months after the last treatment
  Evaluate bone marrow toxicity using absolute neutrophil count

SECONDARY OUTCOMES:
Progression free survival (PFS) | Every 6 months for up to 5 years
  From day 1 of therapy to documented disease progression in CT or MRI as per RECIST criteria
Overall survival (OS) | Up to 5 years
  From start of treatment (cycle 1, day 1) until the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: David Bushnell, MD, Study Chair — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Information will be distributed via clinicaltrials.gov and shared as per the filed NIH data sharing plan
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Typically, after completion of study
Access Criteria: A data sharing agreement will need to be filed for sharing the individual participant data. A contract may be required.

REFERENCES:
- [Background] Bushnell DL, Madsen MT, O'cdorisio T, Menda Y, Muzahir S, Ryan R, O'dorisio MS. Feasibility and advantage of adding (131)I-MIBG to (90)Y-DOTATOC for treatment of patients with advanced stage neuroendocrine tumors. EJNMMI Res. 2014 Dec;4(1):38. doi: 10.1186/s13550-014-0038-2. Epub 2014 Sep 10. PMID 26116109
- [Background] Madsen MT, Bushnell DL, Juweid ME, Menda Y, O'Dorisio MS, O'Dorisio T, Besse IM. Potential increased tumor-dose delivery with combined 131I-MIBG and 90Y-DOTATOC treatment in neuroendocrine tumors: a theoretic model. J Nucl Med. 2006 Apr;47(4):660-7. PMID 16595501
- See also: The website describing the Specialized Programs of Research Excellence in Neuroendocrine Cancers that supports this clinical trial. — https://uihc.org/neuroendocrine-spore-overview